CLINICAL TRIAL: NCT05030116
Title: Comparison of Shenqu Xiaoshi Oral Liquid and Domperidone Suspension in the Treatment of Functional Dyspepsia in Children: a Randomized, Double-blind, Double-simulated, Multi-center Clinical Study
Brief Title: Clinical Trial for 'Shen Qu Xiao Shi' Oral Liquid in the Treatments of Children's Functional Dyspepsia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SQXS20181221
Record Dates: First submitted 2021-08-30; First posted 2021-09-01 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-08

CONDITIONS: Dyspepsia
Keywords: functional dyspepsia; children; Traditional Chinese Medicine
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: Shenqu Xiaoshi oral liquid
- Control Group (Active Comparator)
  Interventions: Drug: Domperidone suspension

INTERVENTIONS:
Drug: Shenqu Xiaoshi oral liquid — Shenqu Xiaoshi oral liquid
  Arms: Experimental group
Drug: Domperidone suspension — Domperidone suspension
  Arms: Control Group

SUMMARY:
With domperidone suspension as the control, the effect of shenqu xiaoshi oral liquid on functional dyspepsia in children was evaluated objectively through multi-center, randomized, double-blind and double-simulation experiment, which alleviated the clinical symptoms, restored and promoted the normal growth and development of children.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 3-14 years, regardless of gender;
2. Meet 1 or more conditions: (1) full after dinner; (2) early full; (3) abdominal pain, and defecation has nothing to do; After appropriate evaluation, symptoms cannot be fully explained by other diseases; Or have other symptoms of dyspepsia, but not caused by other diseases;
3. Have symptoms at least 2 months before diagnosis and at least 4 days per month;
4. During the 2-week leading-in period, no drugs were used to treat infantile anorexia and functional dyspepsia, and good eating habits were established. The patients were fed on time and still had the above-mentioned symptoms of anorexia and functional dyspepsia; The symptom score was 3.
5. The legal guardian of the child should sign the informed consent form. If the child is 10 years old or older, they should sign the informed consent form and agree to participate in the study.

Exclusion Criteria:

1. Anorexia and dyspepsia caused by anorexia or dyspepsia caused by the influence of certain drugs or other confirmed diseases, such as erosive gastritis and gastric ulcer;
2. Children with severe malnutrition;
3. Children with abnormal ecg, liver and kidney functions, nervous system, respiratory system and endocrine system considered by the investigator;
4. Children with mental disorders, dementia and unclear speech;
5. Lactose intolerance or allergy to drug ingredients, or allergy to traditional Chinese medicine;
6. Children who have participated in other clinical trials or are participating in clinical trials of other drugs within 12 weeks; According to the judgment of the researchers, there are other diseases or conditions that reduce the possibility of enrollment or complicate enrollment, such as unstable living environment and inconvenient transportation, which are easy to cause loss and follow-up.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 356 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-23 (Actual)

PRIMARY OUTCOMES:
Total effective rate | Treatment for two weeks

SECONDARY OUTCOMES:
Clinical symptom scores | Treatment for one/two week(s)
Total effective rate | Two weeks after stopping the medication
Food intake | Treatment for one/two week(s) and two weeks after stopping the medication
  Food intake was measured by a scale filling by subjects or their parents. Scores range from 0 to 3. Higher score represents greater reduction in food intake and 0 means unchanged.
weight | Treatment for one/two week(s) and two weeks after stopping the medication
The meal time | Treatment for one/two week(s) and two weeks after stopping the medication
hemoglobin | Treatment for two weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiaotong University School of Medicine Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No